CLINICAL TRIAL: NCT05599373
Title: Optimizing Treatment Protocol of High Frequency Repetitive Transcranial Magnetic Stimulation for Cognitive Deficits and Negative Symptoms in Schizophrenia: an Exploratory Study
Brief Title: Optimal rTMS for Cognitive Deficits and Negative Symptoms in Schizophrenia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Mental Health Center (Other)
Collaborators: Xuhui Mental Health Center (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: XHJW2020KY003
Record Dates: First submitted 2022-10-09; First posted 2022-10-31 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2022-10

CONDITIONS: Schizophrenia; Negative Symptoms in Schizophrenia; Cognitive Impairment; Repetitive Transcranial Magnetic Stimulation; Dorsolateral Prefrontal Cortex
MeSH Terms: conditions — Schizophrenia; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Active rTMS over bilateral dorsolateral prefrontal cortex (Active Comparator): Active rTMS over bilateral dorsolateral prefrontal cortex. Participants will receive up to 20 rTMS sessions within the 4-week treatment period.
  Interventions: Device: Bilateral Active Repetitive transcranial magnetic stimulation (rTMS)
- Active rTMS over left dorsolateral prefrontal cortex (Active Comparator): Active rTMS over left dorsolateral prefrontal cortex and sham rTMS over right dorsolateral prefrontal cortex. Participants will receive up to 20 rTMS sessions within the 4-week treatment period.
  Interventions: Device: Left Active Repetitive transcranial magnetic stimulation (rTMS)
- Sham rTMS over bilateral dorsolateral prefrontal cortex (Sham Comparator): Sham rTMS over bilateral dorsolateral prefrontal cortex. Participants will receive up to 20 rTMS sessions within the 4-week treatment period.
  Interventions: Device: Sham rTMS over bilateral dorsolateral prefrontal cortex

INTERVENTIONS:
Device: Bilateral Active Repetitive transcranial magnetic stimulation (rTMS) — Active treatments with repetitive transcranial magnetic stimulation (rTMS) over bilateral dorsolateral prefrontal cortex (DLPFC) took the form of intermittent theta burst stimulation (iTBS). For iTBS the stimulation parameters were: frequency = triplet 50 Hz bursts, repeated at 5 Hz; train duration = 2 s ON and 8 s OFF, total pulses/session = 600; total number of treatments = 20(5 sessions per week) at 80 % of each side resting motor threshold (MT). The rTMS target was first randomized to the left or right DLPFC, then switched to the opposite side.
  Arms: Active rTMS over bilateral dorsolateral prefrontal cortex
Device: Left Active Repetitive transcranial magnetic stimulation (rTMS) — Active treatments with repetitive transcranial magnetic stimulation (rTMS) over left dorsolateral prefrontal cortex(DLPFC) took the form of intermittent theta burst stimulation (iTBS). For iTBS the stimulation parameters were: frequency = triplet 50 Hz bursts, repeated at 5 Hz; train duration = 2 s ON and 8 s OFF, total pulses/session = 600; total number of treatments = 20(5 sessions per week) at 80 % of left resting motor threshold (MT). Sham rTMS stimulation was delivered over right dorsolateral prefrontal cortex(DLPFC) using the same stimulation parameters, except for using the sham stimulation coil. The rTMS target was first randomized to the left or right DLPFC, then switched to the opposite side.
  Arms: Active rTMS over left dorsolateral prefrontal cortex
Device: Sham rTMS over bilateral dorsolateral prefrontal cortex — Sham rTMS stimulation was delivered over bilateral dorsolateral prefrontal cortex (DLPFC) using the same stimulation parameters, except for using the sham stimulation coil. The rTMS target was first randomized to the left or right DLPFC, then switched to the opposite side.
  Arms: Sham rTMS over bilateral dorsolateral prefrontal cortex

SUMMARY:
Negative symptoms and cognition decline are major challenges in clinical management of schizophrenia. Dorsomedial prefrontal cortex (DLPFC) has been highly involved in the mechanisms of negative symptoms and cognitive symptoms of schizophrenia. However, the effect of repetitive transcranial magnetic stimulation (rTMS) over left or bilateral DLPFC has not yet been well studied. The aim of this study is to describe how the effectiveness of rTMS over different targets for cognitive deficits and negative symptoms in schizophrenia will be evaluated. The study will provide evidence to determine whether a bilateral DLPFC rTMS and is more effective than a left DLPFC rTMS alone to optimize treatment protocol in schizophrenia.

DETAILED DESCRIPTION:
The study will be a randomized, double-blind trial comparing active rTMS over bilateral DLPFC vs. active rTMS over left DLPFC vs. sham rTMS delivered over DLPFC an 4-week treatment period. After assessment and inclusion into the study, participants will be randomized to receive up to 20 sessions of either active rTMS over left DLPFC or bilateral DLPFC or placebo treatments.

ELIGIBILITY:
Inclusion Criteria:

* Met the Diagnostic and Statistical Manual of Mental Disorders, Five Edition (DSM-V) diagnostic criteria for schizophrenia and the diagnosis was verified by an experienced psychiatrist based on the Mini-International Neuropsychiatric Interview (MINI) 7.0 .
* Age between 18 and 60.
* Patients with prominently negative symptoms, which was defined as: PANSS negative subscore≥15 points and one of items N1-N7 scoring≥4.
* All patients were in stable clinical conditions (reduction rate of PANSS score<10% within 4 weeks), stable antipsychotic treatment for at least 4 weeks, and able to provide informed consent.

Exclusion Criteria:

* Any contraindication for rTMS (e.g., intracranial metal, pacemakers, cochlear and intracranial hypertension).
* Unstable clinical condition (e.g., being aggressive and uncooperative).
* Current substance abuse.
* Any other psychiatric diagnosis.
* Significant medical condition including neurological disease, severe cardiovascular, hepatic, renal diseases.
* Previous treatment with modified electric convulsive therapy (MECT) within 3 months before enrollment.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Mean Change From Baseline in Assessment of Negative Symptoms(SANS) Post Treatment | Baseline and 4 weeks
  The Assessment of Negative Symptoms(SANS) is a standardized assessment utilizing a 6-point scale with which the clinician rates the degree to which the severity of the subject's negative symptoms. It consists of 19 items assessing five symptoms of the negative dimension: Affect flattening, alogia, avolition-apathy, anhedonia-asociality, and poor attention.
Mean Change From Baseline in MATRICS Consensus Cognitive Battery Post Treatment | Baseline and 4 weeks
  The MATRICS Consensus Cognitive Batteryis a standardized rating tool to assess the severity of the subject's cognitive symptoms, which consisted of seven domains and the total score: speed of processing, attention/vigilance, working memory, visual learning, verbal learning, reasoning/problem solving, and social cognition.

SECONDARY OUTCOMES:
Mean Change From Baseline in Positive and Negative Syndrome Scale(PANSS)-Negative Symptoms Subscale Post Treatment | Baseline and 4 weeks
  The Positive and Negative Syndrome Scale(PANSS)-Negative Subscale is a valid assessment utilizing a 7 items, 7-point scale with which the clinician rates the degree to which the severity of the subject's negative symptoms.
Mean Change From Baseline in Clinical Global Impression - Severity (CGI-S) Post Treatment | Baseline and 4 weeks
  The Clinical Global Impression - Severity (CGI-S) is a standardized assessment utilizing a single item, 7-point scale with which the clinician rates the severity of the subject's illness at the time of assessment relative to the clinician's past experience with patients who have the same diagnosis.
Mean Change From Baseline in Calgary Depression Scale for Schizophrenia (CDSS) Post Treatment | Baseline and 4 weeks
  Calgary Depression Scale for Schizophrenia (CDSS) is a nine item structures interview scale, in which each item has a four point measure, which has been specifically developed to assess depression in schizophrenics.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Zhan, MD, Principal Investigator — Shanghai Xuhui Mental Health Center
Locations (1):
- Shanghai Xuhui Mental Health Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No